CLINICAL TRIAL: NCT01230957
Title: Safety and Immunogenicity of Different Formulations of a Clostridium Difficile Toxoid Vaccine Administered at Three Different Schedules in Adults Aged 40 to 75 Years at Risk of C. Difficile Infection
Brief Title: Study of Different Formulations of a Clostridium Difficile Toxoid Vaccine Given at Three Different Schedules in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-030-012; UTN: U1111-1114-3917 (Other: WHO)
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Clostridium Difficile Infection; Diarrhea
Keywords: Clostridium difficile infection; Diarrhea; Pseudomembranous colitis; Clostridium Difficile Toxoid Vaccine; ACAM-CDIFF™ vaccine
MeSH Terms: conditions — Clostridium Infections; Diarrhea; Enterocolitis, Pseudomembranous | interventions — Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group 1 (Experimental): Participants will receive a dose Low-dose ACAM-CDIFF™ vaccine with adjuvant on Day 0, 7, and 30, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (Low-dose with adjuvant)
- Group 2 (Experimental): Participants will receive a dose Low-dose ACAM-CDIFF™ vaccine without adjuvant on Day 0, 7, and 30, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (Low-dose without adjuvant)
- Group 3 (Experimental): Participants will receive a dose High-dose ACAM-CDIFF™ vaccine with adjuvant on Day 0, 7, and 30, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant)
- Group 4 (Experimental): Participants will receive a dose High-dose ACAM-CDIFF™ vaccine without adjuvant on Day 0, 7, and 30, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (high-dose without adjuvant)
- Group 5 (Placebo Comparator): Participants will receive a dose Placebo (0.9% normal saline) on Day 0, 7, and 30, respectively.
  Interventions: Biological: Placebo: 0.9% normal saline
- Group 6 (Experimental): Participants will receive a dose of High-dose ACAM-CDIFF™ vaccine with adjuvant on Day 0, 7, and 180, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant)
- Group 7 (Experimental): Participants will receive a dose of High-dose ACAM-CDIFF™ vaccine with adjuvant on Day 0, 30, and 180, respectively.
  Interventions: Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant)

INTERVENTIONS:
Biological: Clostridium difficile toxoids A and B (Low-dose with adjuvant) — 0.5 mL, Intramuscular on Days 0, 7, and 30
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 1
Biological: Clostridium difficile toxoids A and B (Low-dose without adjuvant) — 0.5 mL, Intramuscular on Days 0, 7, and 30
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 2
Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant) — 0.5 mL, Intramuscular on Days 0, 7, and 30
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 3
Biological: Clostridium difficile toxoids A and B (high-dose without adjuvant) — 0.5 mL, Intramuscular on Days 0, 7, and 30
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 4
Biological: Placebo: 0.9% normal saline — 0.5 mL, Intramuscular on Days 0, 7, and 30
  Other Names: 0.9% normal saline
  Arms: Group 5
Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant) — 0.5 mL, Intramuscular on Days 0, 7, and 180
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 6
Biological: Clostridium difficile toxoids A and B (high-dose with adjuvant) — 0.5 mL, Intramuscular on Days 0, 30, and 180
  Other Names: ACAM-CDIFF™ vaccine
  Arms: Group 7

SUMMARY:
This study will further evaluate the ACAM-CDIFF™ vaccine in a population of middle-aged to elderly individuals at risk of exposure to Clostridium difficile because of impending hospitalization or residence in a care facility.

Primary Objectives:

* To describe the safety profile of subjects in each of the study groups.
* To describe the immune responses elicited by toxoid A and toxoid B of subjects in each of the study groups.

Observational Objective:

* To describe the occurrence of first-time Clostridium difficile infection (CDI) episodes.

DETAILED DESCRIPTION:
Participants will receive 3 doses of either one of 4 different formulations of ACAM-CDIFF™ vaccine or placebo, on one of 3 different schedules. The trial will have 2 stages. Stage I will test 4 different formulations of ACAM-CDIFF™ vaccine. Stage II will explore different vaccination schedules using one of these formulations.

Participants will be followed up for safety and immunogenicity; stool samples will also be provided in case of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 75 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination
* At risk for developing Clostridium difficile infection during the trial because of impending elective surgery or hospitalization within 60 days of enrollment, or current or impending residence in a long-term care facility or rehabilitation facility.

Exclusion Criteria:

* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for influenza (seasonal or pandemic) and pneumococcal vaccine
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination, except for influenza (seasonal or pandemic) and pneumococcal vaccines
* Previous vaccination against Clostridium difficile with either the trial vaccine or another vaccine
* Current or prior Clostridium difficile infection (CDI) episode
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C
* Anticipated or current receipt of kidney dialysis treatment
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as a study site employee who is involved in the protocol and may have direct access to trial-related data
* Subjects who have any history of intestinal diverticular bleeding
* Subjects who have had surgery within the past three months for gastrointestinal (GI) malignancy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Information concerning the safety profile in terms of solicited and unsolicited reactions in participants following vaccination with ACAM-CDIFF™ Vaccine. | 6 days after each vaccination and up to 6 months post-vaccination 3
Serum antitoxin IgG concentrations to Clostridium difficile toxins A and B in participants vaccinated with ACAM-CDIFF™. | Up to 6 months post-vaccination 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (28):
- United States (28):
  - Redding, California
  - Bristol, Connecticut
  - Stamford, Connecticut
  - Clearwater, Florida
  - Coral Gables, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Newton, Kansas
  - Brockton, Massachusetts
  - Troy, Michigan
  - Neptune City, New Jersey
  - Binghamton, New York
  - Endwell, New York
  - Cary, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Centerville, Ohio
  - Pittsburgh, Pennsylvania
  - Uniontown, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Williamsburg, Virginia
  - Marshfield, Wisconsin

REFERENCES:
- [Result] de Bruyn G, Saleh J, Workman D, Pollak R, Elinoff V, Fraser NJ, Lefebvre G, Martens M, Mills RE, Nathan R, Trevino M, van Cleeff M, Foglia G, Ozol-Godfrey A, Patel DM, Pietrobon PJ, Gesser R; H-030-012 Clinical Investigator Study Team. Defining the optimal formulation and schedule of a candidate toxoid vaccine against Clostridium difficile infection: A randomized Phase 2 clinical trial. Vaccine. 2016 Apr 27;34(19):2170-8. doi: 10.1016/j.vaccine.2016.03.028. Epub 2016 Mar 21. PMID 27013431
- [Derived] Small RD, Ozol-Godfrey A, Yan L. On the use of nonparametric tests for comparing immunological Reverse Cumulative distribution curves (RCDCs). Vaccine. 2019 Oct 16;37(44):6737-6742. doi: 10.1016/j.vaccine.2019.09.007. Epub 2019 Sep 16. PMID 31537446